CLINICAL TRIAL: NCT06426966
Title: Comparative Efficacy of Gymnema Sylvestre vs Berberine in the Clinical Outcomes and Gene Expression of Adipokines in Patients With Exogenous Obesity
Brief Title: Gymnema Sylvestre vs Berberine in Obesity Gene Expression of Adipokines
Acronym: GS VS BBR A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Polytechnic Institute, Mexico (Other)
Collaborators: Instituto Nacional de Pediatria (Unknown)
Responsible Party: Principal Investigator, Cindy Rodríguez Bandala, PhD, National Polytechnic Institute, Mexico
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESM.CE-01/7-12-2015; 20170253 (Other: Instituto Politécnico Nacional México)
Record Dates: First submitted 2024-05-15; First posted 2024-05-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Diabetes Mellitus; Obesity
Keywords: Diabetes; Gymnema sylvestre; Berberine; adipokines; obesity
MeSH Terms: conditions — Diabetes Mellitus; Obesity | interventions — Berberine; Gurmarin protein, Gymnema sylvestre

STUDY DESIGN:
Intervention Model Description: Comparative, quasi-experimental
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gymnema sylvestre (Experimental): Patients who present Obesity administrated with Gymnema sylvestre. At a dose of two 200 mg capsules before breakfast
  Interventions: Dietary Supplement: Gymnema sylvestre
- Berberine (Experimental): Patients who present Obesity administrated with Berberine 500 mg tablet three times a day before each meal
  Interventions: Dietary Supplement: Berberine

INTERVENTIONS:
Dietary Supplement: Berberine — Berberine is an alkaloid derived from plants native to China called Rhizoma coptidis, Cortex phellodendrine and Hydrastis canadensis. These plants are used in the treatment of infectious diarrhea, inflammation, DM2, non-alcoholic fatty liver disease, dyslipidemias, cardiovascular diseases, and obesity. They have been shown to improve insulin sensitivity and stimulate glucose uptake through the activation of AMP-activated protein kinase (AMPK)
  Arms: Berberine
Dietary Supplement: Gymnema sylvestre — Gymnema sylvestre also known as "meshashringi", is a plant from central and southern India. The leaf extract has been used as a laxative, diuretic, and cough suppressant; Likewise, it has antimicrobial, antihypercholesterolemic, and hepatoprotective activities. It is associated with antioxidant properties . Its adjuvant effect has been reported in the therapy of type 2 diabetes, revealing how its active compounds can influence glucose regulation and improve insulin sensitivity.
  Arms: Gymnema sylvestre

SUMMARY:
Obesity is a disease that affects a large part of the world's population and is a risk factor for the development of metabolic, cardiovascular, oncological, and neurodegenerative diseases. Treatments with Gymnema Sylvestre (GS) and Berberine (BBR) have been studied in metabolic diseases such as obesity and type 2 diabetes mellitus (DM2), and have gained importance in recent years, however, questions remain regarding their comparative effect on biochemical parameters, body composition and gene expression of adipokines. Methodology. We carried out a comparative study in 50 adult Mexican patients with a diagnosis of Obesity. Two groups of patients were formed: A. Treated with GS and B. Treated with BBR. Baseline and final measurements were determined 3 months after treatment. Biochemical and body composition parameters were evaluated and the gene expression of Resistin (Res), Omentin (Om), Visfatin (Vis) and Apelin (Ap) was determined, as well as safety parameters.

DETAILED DESCRIPTION:
Trial oversight A comparative, descriptive, observational, longitudinal, and prospective analysis study was carried out in the Comprehensive Obesity and Overweight Care Program at the Higher School of Medicine. This study was carried out in full accordance with good clinical practice guidelines and the Declaration of Helsinki. The study was registered with the Research and Ethics Committee of the Higher School of Medicine (ESM.CE-01/7-12-2015). All patients signed the informed consent, and the information was protected through a confidentiality letter.

Patients We included 50 Mexican patients of both sexes, of the over 18 years of age, with a body mass index (BMI) greater than 30 KG(kilogram)/M2 (obesity grade I, II and III), without a previous diagnosis of diabetes mellitus, but with at least two risk factors for the disease (history of parents or siblings, over 40 years of age, sedentary lifestyle habits, controlled arterial hypertension, fasting blood glucose < 126 mg/dL or glycated hemoglobin < 6.5%). Key exclusion criteria included (i) pregnant patients, (ii) diabetics, and (iii) patients with allergic reaction to any components of the supplements. The first study group, group A (25 patients) was treated with GS at a dose of two 200 mg capsules before breakfast, while in the second group, group B (25 patients) were treated with BBR at dose of one 500 mg tablet three times a day before each meal. In both groups, the treatment lasted 3 months.

Trial procedures and outcomes Anthropometric, physiological, and biochemical parameters were measured in two sessions, before and after treatment. The anthropometric measurements were body weight, height, waist, and hip circumference, in addition to body analysis using the Inbody 770. As a physiological measure, only blood pressure was considered using WelchAllyn brand anomanometers with cuff for obese patients. Regarding biochemical parameters, fasting glucose, lipid profile (total cholesterol, triglycerides, HDL, LDL), basal insulin and HbA1c were measured. Adherence to treatment and the presence of adverse effects was recorded using a log that indicated the time at which the tablets were ingested and whether they had any adverse effects that day.

Additionally, whole blood samples were taken from 50 patients, 25 had received treatment with GS (group A) and 25 received treatment with BBR (group B). The extraction of tRNA(transfer ribonucleic acid) was carried out using the TRIzol®Reagent technique, which consists of a mixture of guanidine isocyanate and phenol-chloroform. Once the total RNA was isolated, it was suspended in RNase-free water to avoid possible degradation of the sample before proceeding with reverse transcription. The extraction and integrity of the tRNA was verified by means of agarose gel electrophoresis. The final purity of the samples was calculated based on the absorbance obtained with a measurement at 260-280. cDNA(complementary DNA) amplification was performed using the "First Strand cDNA transcription" synthesis kit for rtPCR from Roche. A real-time polymerase chain reaction (RT-PCR) procedure was performed to determine the relative expression of the mRNA(messenger ribonucleic acid) of the genes studied, using probes from the human transcriptome library (Human Universal Probe Library), a LightCycler nano thermocycler and a TaqMan type reaction mixture, all from the Roche Diagnostics brand (Roche Diagnostics GmbH(Gesellschaft mit beschränkter Haftung), Mannheim, Germany). The oligo sequences of the primers (sense and antisense) were designed with ProbeFinder software (Apelin, NM_017413.4, F, 5´ gaa agt ggg gga tgg cta ag 3´, R, 5´ ccc acc cac tac cct ctt ct 3´, Omentin, NM_017625.2, F, 5´ tga ggg tca ccg gat gta ac 3´, R, 5´ gga ctg gcc tct gga aag ta 3´, Resistin, NM_001193374.1, F, 5´ cca ccg aga ggg atg aaa g 3´, R, 5´ ttc ttc cat gga gca cag g 3´ and Visfatin, NM_005746.2, F, 5´ aag gga tgg aac tac att ctt gag 3´, R, 5´ ctg tgt ttt cca ccg tga ag 3'. The reaction mix was prepared according to the manufacturer's protocol. Each sample was analyzed in duplicate, and the data obtained were analyzed with the LightCycler nano software.

Statistical analysis The distribution of the quantitative data was performed by Shapiro Wilk. The comparison of frequencies was carried out with X2, while the comparison of basal means between groups was performed with Student's t-test. Final means were compared with Student's t-test when no statistical differences were found in basal comparison, while in the parameters with significant differences in the basal measurement, a covariate adjustment (repeated measures ANOVA) and the Bonferroni test were applied to compare the final means between groups. Self-controlled analysis was performed with paired t test. Analyses were performed with GraphPad Prism software, version 8.0.0 for Windows (GraphPad Software, San Diego, CA, USA), and SPSS software, version 19 (IBM Corp. Released 2015. IBM SPSS Statistics for Windows, Version 19.0. Armonk, NY(New York), USA: IBM Corp). A value of p<0.05 was considered as statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Mexican patients of both sexes, of the over 18 years of age, with a body mass index (BMI) greater than 30 KG/M2 (obesity grade I, II and III), without a previous diagnosis of diabetes mellitus, but with at least two risk factors for the disease (history of parents or siblings, over 40 years of age, sedentary lifestyle habits, controlled arterial hypertension, fasting blood glucose < 126 mg/dL or glycated hemoglobin < 6.5%)

Exclusion Criteria:

* pregnant patients,
* diabetics,
* patients with allergic reaction to any components of the supplements

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Body weight | 3 months
  Body weight
height | 3 months
  height
waist | 3 months
  waist long
hip circumference | 3 months
  hip circumference

SECONDARY OUTCOMES:
blood pressure | 3 months
  blood pressure

IPD SHARING:
Plan to Share IPD: No
Publication of the article in a JCR journal

REFERENCES:
- [Background] Zhang X, Ha S, Lau HC, Yu J. Excess body weight: Novel insights into its roles in obesity comorbidities. Semin Cancer Biol. 2023 Jul;92:16-27. doi: 10.1016/j.semcancer.2023.03.008. Epub 2023 Mar 24. PMID 36965839
- [Background] Zwick RK, Guerrero-Juarez CF, Horsley V, Plikus MV. Anatomical, Physiological, and Functional Diversity of Adipose Tissue. Cell Metab. 2018 Jan 9;27(1):68-83. doi: 10.1016/j.cmet.2017.12.002. PMID 29320711
- [Background] Recinella L, Orlando G, Ferrante C, Chiavaroli A, Brunetti L, Leone S. Adipokines: New Potential Therapeutic Target for Obesity and Metabolic, Rheumatic, and Cardiovascular Diseases. Front Physiol. 2020 Oct 30;11:578966. doi: 10.3389/fphys.2020.578966. eCollection 2020. PMID 33192583
- [Background] Steppan CM, Bailey ST, Bhat S, Brown EJ, Banerjee RR, Wright CM, Patel HR, Ahima RS, Lazar MA. The hormone resistin links obesity to diabetes. Nature. 2001 Jan 18;409(6818):307-12. doi: 10.1038/35053000. PMID 11201732
- [Background] Revollo JR, Korner A, Mills KF, Satoh A, Wang T, Garten A, Dasgupta B, Sasaki Y, Wolberger C, Townsend RR, Milbrandt J, Kiess W, Imai S. Nampt/PBEF/Visfatin regulates insulin secretion in beta cells as a systemic NAD biosynthetic enzyme. Cell Metab. 2007 Nov;6(5):363-75. doi: 10.1016/j.cmet.2007.09.003. PMID 17983582
- [Background] Dakroub A, A Nasser S, Younis N, Bhagani H, Al-Dhaheri Y, Pintus G, Eid AA, El-Yazbi AF, Eid AH. Visfatin: A Possible Role in Cardiovasculo-Metabolic Disorders. Cells. 2020 Nov 9;9(11):2444. doi: 10.3390/cells9112444. PMID 33182523
- [Background] Ugur K, Erman F, Turkoglu S, Aydin Y, Aksoy A, Lale A, Karagoz ZK, Ugur I, Akkoc RF, Yalniz M. Asprosin, visfatin and subfatin as new biomarkers of obesity and metabolic syndrome. Eur Rev Med Pharmacol Sci. 2022 Mar;26(6):2124-2133. doi: 10.26355/eurrev_202203_28360. PMID 35363362
- [Background] Huang J, Kang S, Park SJ, Im DS. Apelin protects against liver X receptor-mediated steatosis through AMPK and PPARalpha in human and mouse hepatocytes. Cell Signal. 2017 Nov;39:84-94. doi: 10.1016/j.cellsig.2017.08.003. Epub 2017 Aug 15. PMID 28821440
- [Background] Li C, Cheng H, Adhikari BK, Wang S, Yang N, Liu W, Sun J, Wang Y. The Role of Apelin-APJ System in Diabetes and Obesity. Front Endocrinol (Lausanne). 2022 Mar 9;13:820002. doi: 10.3389/fendo.2022.820002. eCollection 2022. PMID 35355561
- [Background] Sperling M, Grzelak T, Pelczynska M, Bogdanski P, Formanowicz D, Czyzewska K. Association of Serum Omentin-1 Concentration with the Content of Adipose Tissue and Glucose Tolerance in Subjects with Central Obesity. Biomedicines. 2023 Jan 24;11(2):331. doi: 10.3390/biomedicines11020331. PMID 36830868
- See also: World Health Organization: WHO. — https://www.who.int/es/news-room/fact-sheets/detail/obesity-and-overweight